CLINICAL TRIAL: NCT06424496
Title: Effect of Targeted Health Education Program on Nurses' Awareness About Postpartum Depression
Acronym: PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rasha Saad, Assistant professor of Epidemiology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Nurses' Awareness About PPD
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Quazi-Experimental study (pre/post design).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An intervention study (a quasi-experimental design) (Other): An intervention study (a quasi-experimental design)pre&post
  Interventions: Other: Effect of Targeted Health Education Program on Nurses' Awareness About Postpartum Depression

INTERVENTIONS:
Other: Effect of Targeted Health Education Program on Nurses' Awareness About Postpartum Depression — Quazi-Experimental study (pre/post design) to assess the Effect of Targeted Health Education Program on Nurses' Awareness About Postpartum Depression
  Other Names: Quazi-Experimental study (pre/post design).

SUMMARY:
To assess nurses' knowledge of PPD at Ain Shams University Maternity Hospital and measure their knowledge level after an educational program on postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a serious mental illness that involves the brain and affects behavior and physical health of women after childbirth . Multiple factors may influence PPD, such as lack of support, interpersonal events, withdrawal of hormones after delivery, psychosocial stressors, psychological stressors, personality, environment, and ineffective adaptation.

Symptoms of PPD may include feeling restless or moody, feeling sad, crying a lot, having thoughts about hurting the baby or yourself, not feeling connected to the baby, having no energy or motivation, eating, or sleeping too little or too much, feeling worthless and guilty, losing interest or pleasure in activities, and withdrawing from friends and family .

PPD is one of the most important health problems due to its prevalence; 10-15% . and serious negative mother-baby outcomes. PPD affects the health of mothers and their newborns and is associated with long-term psychological and socioeconomic implications .

As the knowledge affects attitudes and practices of people, nurses' knowledge can affect profoundly women after birth specially regarding PPD .

In an American web-based study , nurses' self-efficacy about PPD was associated to their knowledge . In another American electronic survey of 372 nurses, 95% reported an association between post-partum education and mortality and 72% reported that it is their responsibility to provide education to mothers .

In a Ghanaian study, nurses had good knowledge about PPD but poor knowledge about screening and management . In a Kazakh study, 90% of nurses didn't attend training courses on PPD ).

Furthermore, in a Malaysian study, 44.4 % of participants were below than median total knowledge score and only 25.9% practiced screening. In a Saudi study, the confidence of nurses and midwives to educate women about PPD was associated with their knowledge. In a Turkish study, 84.4 % of nurses had little knowledge and 75.5% reported that psychological service for evaluating mothers wasn't offered.

PPD can have devastating effects on women, their infants, and families associated with lower levels of bonding and reduced breastfeeding initiation and duration. Consequently, women experiencing PPD may cause harm to their baby, themselves, or others.

As, nurses in Maternity Hospitals are poised to play a pivotal role in the early identification and prompt treatment of PPD, assessing their knowledge is very important. To date, according to our knowledge, there is no previous study in Egypt assessing the nurses' knowledge about PPD, therefore the present study will be conducted to compare their knowledge regarding PPD before and after the health education program.

ELIGIBILITY:
Inclusion Criteria:

* Nurses at Ain Shams University Maternity Hospital

Exclusion Criteria:

none

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
To measure the mean change in the nurses' knowledge score after applying the health education program about postpartum depression | one month
  Evaluate the effect of the targeted health education program on nurses' knowledge score using a self-administer questionnaire consisting of 28 items covering main issues regarding prevalence risk factors, symptoms, and treatment of PPD. The answer to each question had two options (true or false). The total score ranges from 0-28

CONTACTS AND LOCATIONS:
Overall Officials: rasha saad Hussein, MD, Principal Investigator — Faculty of medicine Ain shams univrsity
Locations (1):
- faculty of medicine Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No